CLINICAL TRIAL: NCT04816526
Title: Phase 2 Study of Descartes-08 Consolidation Treatment in Patients With High-Risk Multiple Myeloma Who Have Residual Disease After Induction Therapy
Brief Title: Descartes-08 Consolidation Treatment in Patients With High-Risk Multiple Myeloma High-Risk Multiple Myeloma Who Have Residual Disease After Induction Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-08-B
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Myeloma Multiple
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Descartes 08 (Experimental)
  Interventions: Biological: Descartes 08

INTERVENTIONS:
Biological: Descartes 08 — Car T-cells

SUMMARY:
To assess Minimal Residual Disease (MRD)-negative Complete Response (sCR) rate after consolidation treatment with Descartes-08 in patients with high-risk myeloma who have residual disease following induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older at the time of enrollment
* High-risk multiple myeloma patients who complete pre-transplant induction treatment anti- myeloma drug combination (minimum 2 drugs).

Exclusion Criteria:

* Patients who are pregnant or lactating.
* Patients who have any active and uncontrolled infection. No blood cultures are necessary unless clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California Irvine, Orange, California
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Descartes 08: Six IV infusions of Descartes-08 on Days 1, 4, 11, 15, 18 at 30X10^6 cells/kg.
Period: Overall Study
Arm/Group | Descartes 08
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Descartes 08
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10
  Turkey | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Stringent Complete Response
Description: Per IMWG 2016 Response Criteria Summary sCR: Complete response (CR) plus a normal free light chain ratio and no clonal cells in bone marrow (by immunohistochemistry). The FLC ratio must be Kappa/Lambda ≤ 4:1 or ≥ 1:2 after counting at least 100 plasma cells. CR: Negative immunofixation in serum and urine, disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow. VGPR: Serum M-protein detectable by immunofixation (not on electrophoresis) or a ≥ 90% reduction in M-protein, with urine M-protein <100 mg/24 hours. PR: ≥ 50% reduction in serum M-protein and a ≥ 90% reduction in 24-hour urinary M-protein (or to <200 mg/24 hours). If M-protein is unmeasurable, a ≥ 50% decrease in the difference between involved and uninvolved FLC levels is required. If both M-protein and serum-free light chains are unmeasurable, a ≥ 50% reduction in plasma cells is necessary, provided baseline plasma-cell percentage in bone marrow was ≥ 30%. Overall Response (OR): CR+VGPR+PR
Time Frame: 8 months
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Descartes 08
Number analyzed (Participants) | 13
Participants | 7

ADVERSE EVENTS:
Time Frame: Through study completion, median follow up of 5.6 months with a range of 2-11 months.
Arm/Group | Descartes 08
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Descartes 08 (N=13)
Fever (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Descartes 08 (N=13)
Fever (Immune system disorders) | 5 (8)
Chills (Immune system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04816526/Prot_SAP_001.pdf